CLINICAL TRIAL: NCT00696709
Title: A Phase I, Double-Blind, Randomized, Placebo-Controlled Clinical Trial to Evaluate the Safety, Tolerability and Immunogenicity of V212 in Healthy Adults
Brief Title: A Study to Test the Safety and Antibody Response of V212 in Healthy Adults (V212-004)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V212-004; V212-004 (Other: Merck)
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Results first posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-10

CONDITIONS: Herpes Zoster
Keywords: Herpes Zoster (Shingles)
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part 1: Heat-treated Varicella-Zoster Virus (VZV) Vaccine (Experimental): Participants received an 0.65 mL subcutaneous injection of heat-treated varicella zoster virus (VZV) vaccine A; 4-dose regimen administered ~30 days apart.
  Interventions: Biological: Comparator: V212
- Part 1: Gamma- Irradiated VZV Vaccine A (Experimental): Participants received an 0.65 mL subcutaneous injection of alternative inactivation method VZV vaccine A; 4-dose regimen administered ~30 days apart.
  Interventions: Biological: Comparator: V212
- Part 1: Placebo (Placebo Comparator): Participants received a 4-dose placebo regimen administered ~30 days apart.
  Interventions: Biological: Comparator: Placebo
- Part 2: Gamma- Irradiated VZV Vaccine B (Experimental): Participants received an 0.65 mL subcutaneous injection of alternative inactivation method VZV vaccine B; 4-dose regimen administered ~30 days apart.
  Interventions: Biological: Comparator: V212
- Part 2: Gamma- Irradiated VZV Vaccine C (Experimental): Participants received an 0.65 mL subcutaneous injection of alternative inactivation method VZV vaccine C; 4-dose regimen administered ~30 days apart.
  Interventions: Biological: Comparator: V212

INTERVENTIONS:
Biological: Comparator: V212 — 0.65 mL subcutaneous injection of heat-treated Varicella zoster virus (VZV) vaccine or alternative inactivation method VZV vaccine A, B, C; 4-dose regimen administered ~30 days apart
  Arms: Part 1: Gamma- Irradiated VZV Vaccine A; Part 1: Heat-treated Varicella-Zoster Virus (VZV) Vaccine; Part 2: Gamma- Irradiated VZV Vaccine B; Part 2: Gamma- Irradiated VZV Vaccine C
Biological: Comparator: Placebo — Placebo; 4-dose regimen administered ~30 days apart.
  Arms: Part 1: Placebo

SUMMARY:
The purpose of this study was to assess the safety and tolerability of gamma-irradiated varicella-zoster virus (VZV) vaccine A (Part 1) and gamma-irradiated VZV vaccine B and C (Part 2) and to determine if they were immunogenic when administered to healthy individuals, as measured by VZV-specific antibody responses by glycoprotein enzyme-linked immunosorbent assay (gpELISA). The primary hypothesis was that gamma-irradiated VZV vaccine A (Part 1) and gamma-irradiated VZV vaccine B and C (Part 2) would elicit an acceptable VZV-specific immune response. The secondary hypothesis for Part 1 of the study was that heat-treated VZV vaccine would elicit an acceptable VZV-specific immune response.

ELIGIBILITY:
Inclusion Criteria:

* Must be 50 to 59 years of age
* No fever on vaccination days
* Must have had chickenpox or lived in an area where the chickenpox virus is prevalent for 30 or more years
* Females of child-bearing potential must use acceptable forms of birth control

Exclusion Criteria:

* Prior history of shingles
* Prior receipt of any chickenpox or shingles vaccine
* Pregnant or breastfeeding
* Received or expect to receive a live virus vaccine (such as measles, mumps, rubella) from 4 weeks before the first visit through the last visit
* Received or expect to receive an inactivated vaccine (such as tetanus or pneumonia) from 7 days before the first visit through the last visit
* Received immunoglobulin or blood products
* Receiving treatment that may weaken the immune system
* Have an immune system disorder

Ages: 50 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 290 (Actual)
Dates: Start 2008-12-12 (Actual); Primary Completion 2009-11-16 (Actual); Study Completion 2009-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed in 2 parts - Part 1 and Part 2, with a total of 160 participants.
Pre-assignment Details: In Part 1, all participants received heat-treated varicella zoster virus (VZV) vaccine, gamma-irradiated VZV vaccine A or placebo administered as a 4-dose regimen approximately every 30 days. In Part 2, all participants received either gamma-irradiated VZV vaccine B or C administered as a 4-dose regimen approximately every 30 days.
Groups:
- Part 1: Heat-treated Varicella-Zoster Virus (VZV) Vaccine: Participants received an 0.65 mL subcutaneous injection of heat-treated VZV vaccine A; 4-dose regimen administered ~30 days apart.
- Part 1: Gamma-Irradiated VZV Vaccine A: Participants received an 0.65 mL subcutaneous injection of alternative inactivation method VZV vaccine A; 4-dose regimen administered ~30 days apart.
- Part 2: Gamma-Irradiated VZV Vaccine B: Participants received an 0.65 mL subcutaneous injection of alternative inactivation method VZV vaccine B; 4-dose regimen administered ~30 days apart.
- Part 2: Gamma-Irradiated VZV Vaccine C: Participants received an 0.65 mL subcutaneous injection of alternative inactivation method VZV vaccine C; 4-dose regimen administered ~30 days apart.
Period: Overall Study
Arm/Group | Part 1: Heat-treated Varicella-Zoster Virus (VZV) Vaccine | Part 1: Gamma-Irradiated VZV Vaccine A | Part 1: Placebo | Part 2: Gamma-Irradiated VZV Vaccine B | Part 2: Gamma-Irradiated VZV Vaccine C
Started | 65 | 63 | 33 | 64 | 65
Vaccination 1 (Day 1) | 65 | 63 | 32 | 64 | 65
Vaccination 2 (~Day 30) | 64 | 60 | 32 | 61 | 64
Vaccination 3 (~Day 60) | 64 | 60 | 32 | 59 | 63
Vaccination 4 (~Day 90) | 62 | 60 | 32 | 59 | 63
Completed | 62 | 60 | 32 | 59 | 62
Not Completed | 3 | 3 | 1 | 5 | 3
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 4 | 3
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Heat-treated Varicella-Zoster Virus (VZV) Vaccine | Part 1: Gamma-Irradiated VZV Vaccine A | Part 1: Placebo | Part 2: Gamma-Irradiated VZV Vaccine B | Part 2: Gamma-Irradiated VZV Vaccine C | Total
Number analyzed (Participants) | 65 | 63 | 33 | 64 | 65 | 290
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.0 (2.6) | 54.0 (2.5) | 54.0 (2.9) | 53.9 (3.0) | 54.6 (3.1) | 54.1 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 45 | 25 | 42 | 37 | 193
  Male | 21 | 18 | 8 | 22 | 28 | 97

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Geometric Mean Fold Rise of the Varicella-Zoster Virus (VZV)-Specific Immune Responses Measured by Glycoprotein Enzyme-Linked Immunosorbent Assay in Gamma-Irradiated VZV Vaccine A Recipients
Description: Serum samples were tested for antibody response using a glycoprotein enzyme-linked immunosorbent assay (gpELISA) in gamma-irradiated VZV vaccine A recipients. The geometric mean fold rise (GMFR) is the response at approximately 28 days postdose 4 / response predose on Day 1. This outcome measure applied only to participants who received VZV vaccine A; heat-treated VZV vaccine and placebo participants were not assessed for this outcome.
Time Frame: Baseline and ~28 days Postdose 4 (~Day 118)
Population: The analysis population included all gamma-irradiated VZV vaccine A participants who received all 4 vaccinations with no protocol deviations; heat-treated VZV vaccine, vaccine B, vaccine C and placebo participants were not assessed for this outcome.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Part 1: Gamma- Irradiated VZV Vaccine A
Number analyzed (Participants) | 59
Ratio | 2.18 [1.82 to 2.61]
Statistical Analysis 1: Comparison: Part 1: Gamma- Irradiated VZV Vaccine A; Test type: Other; p < 0.0001, Longitudinal regression (LR) — The statistical criterion for significance requires that the lower bound of the 2-sided 95% confidence interval of the geometric mean fold rise in vaccine recipients is >1.0; Calculated based on LR model (adjusting for pre-vaccination immunogenicity level and incomplete data) with visit as covariate

2. Primary Outcome: Part 2: Geometric Mean Fold Rise of the VZV-Specific Immune Responses Measured by gpELISA in Gamma-Irradiated VZV Vaccine B Recipients
Description: Serum samples were tested for antibody response using gpELISA in gamma-irradiated VZV vaccine B recipients. The GMFR is the response at approximately 28 days postdose 4 / response predose on Day 1.
Time Frame: Baseline and ~28 days Postdose 4 (~Day 118)
Population: The analysis population included all gamma-irradiated VZV vaccine B participants who received all 4 vaccinations with no protocol deviations; heat-treated VZV vaccine, vaccine A, vaccine C and placebo participants were not assessed for this outcome.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Part 2: Gamma-Irradiated VZV Vaccine B
Number analyzed (Participants) | 59
Ratio | 1.90 [1.57 to 2.29]
Statistical Analysis 1: Comparison: Part 2: Gamma-Irradiated VZV Vaccine B; Test type: Other; p < 0.0001, Longitudinal regression (LR) — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

3. Primary Outcome: Part 2: Geometric Mean Fold Rise of the VZV-Specific Immune Responses Measured by gpELISA in Gamma-Irradiated VZV Vaccine C Recipients
Description: Serum samples were tested for antibody response using gpELISA in gamma-irradiated VZV vaccine C recipients. The GMFR is the response at approximately 28 days postdose 4 / response predose on Day 1.
Time Frame: Baseline and ~28 days Postdose 4 (~Day 118)
Population: The analysis population included all gamma-irradiated VZV vaccine C participants who received all 4 vaccinations and had no protocol deviations; heat-treated VZV vaccine, vaccine A, vaccine B and placebo participants were not assessed for this outcome.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Groups:
- Part 2: Gamma-Irradiated VZV Vaccine C: Participants received an 0.65 mL subcutaneous injection of heat-treated varicella zoster virus (VZV) vaccine or alternative inactivation method VZV vaccine A, B, C; 4-dose regimen administered ~30 days apart.
Arm/Group | Part 2: Gamma-Irradiated VZV Vaccine C
Number analyzed (Participants) | 63
Ratio | 1.58 [1.35 to 1.84]
Statistical Analysis 1: Comparison: Part 2: Gamma-Irradiated VZV Vaccine C; Test type: Other; p < 0.0001, Longitudinal regression (LR) — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Part 1: Geometric Mean Fold Rise of the Heat-Treated VZV-Specific Immune Responses Measured by gpELISA
Description: Serum samples were tested for antibody response using gpELISA in heat-treated VZV vaccine recipients. The GMFR is the response at approximately 28 days postdose 4 / response predose on Day 1.
Time Frame: Baseline and ~28 days Postdose 4 (~Day 118)
Population: The analysis population included all heat-treated VZV vaccine participants who received all 4 vaccinations and had no protocol deviations; vaccine A, vaccine B, vaccine C and placebo participants were not assessed for this outcome.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Part 1: Heat-treated Varicella-Zoster Virus (VZV) Vaccine
Number analyzed (Participants) | 62
Ratio | 2.10 [1.78 to 2.48]
Statistical Analysis 1: Comparison: Part 1: Heat-treated Varicella-Zoster Virus (VZV) Vaccine; Test type: Other — The statistical criterion for significance requires that the lower bound of the 2-sided 95% confidence interval of the geometric mean fold rise in vaccine recipients is >1.0; p < 0.0001, Longitudinal data analysis (LDA); LDA with log-transformed VZV responses at each visit as response variables and visit as covariate

5. Primary Outcome: Percentage of Participants With a Serious Adverse Event
Description: A serious adverse event (SAE) is defined as an adverse event that resulted in death, was life threatening, resulted in persistent or significant disability or incapacity, resulted in or prolonged a hospitalization, or is a congenital anomaly or birth defect. The percentage of participants with one or more SAEs was assessed.
Time Frame: Up to ~28 days Postdose 4 (Up to ~118 days)
Population: The analysis population included all participants who received at least one dose of vaccine and who had any safety follow-up based on the actual vaccination received. Participants were excluded if they received an incorrect vaccination.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1: Heat-treated Varicella-Zoster Virus (VZV) Vaccine | Part 1: Gamma-Irradiated VZV Vaccine A | Part 1: Placebo | Part 2: Gamma-Irradiated VZV Vaccine B | Part 2: Gamma-Irradiated VZV Vaccine C
Number analyzed (Participants) | 64 | 61 | 32 | 63 | 65
Percentage of Participants | 0.0 | 1.6 | 0.0 | 1.6 | 0.0
Statistical Analysis 1: Comparison: Part 1: Heat-treated Varicella-Zoster Virus (VZV) Vaccine vs Part 1: Placebo; Test type: Other; Difference in Percentage = 0.0, 95% CI 2-sided [-10.8 to 5.7] — Miettinen & Nurminen
Statistical Analysis 2: Comparison: Part 1: Gamma-Irradiated VZV Vaccine A vs Part 1: Placebo; Test type: Other; Difference in Percentage = 1.6, 95% CI 2-sided [-9.2 to 8.8] — Miettinen & Nurminen

6. Primary Outcome: Percentage of Participants With an Injection-Site Adverse Event Prompted on the Vaccination Report Card
Description: An adverse event (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the study vaccine. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an AE. Vaccination Report Card (VRC)-prompted injection-site AEs included redness, swelling, and pain/tenderness/soreness. The percentage of participants with one or more VRC prompted injection-site AE was assessed with incidence > 0% in one or more vaccination groups.
Time Frame: Up to Day 5 post any vaccination (Up to ~5 days)
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1: Heat-treated Varicella-Zoster Virus (VZV) Vaccine | Part 1: Gamma-Irradiated VZV Vaccine A | Part 1: Placebo | Part 2: Gamma-Irradiated VZV Vaccine B | Part 2: Gamma-Irradiated VZV Vaccine C
Number analyzed (Participants) | 64 | 61 | 32 | 63 | 65
Percentage of Participants | 57.8 | 62.3 | 21.9 | 63.5 | 50.8
Statistical Analysis 1: Comparison: Part 1: Heat-treated Varicella-Zoster Virus (VZV) Vaccine vs Part 1: Placebo; Test type: Other; p < 0.001, Miettinen & Nurminen; Difference in Percentage = 35.9, 95% CI 2-sided [15.2 to 52.6]
Statistical Analysis 2: Comparison: Part 1: Gamma-Irradiated VZV Vaccine A vs Part 1: Placebo; Test type: Other; p < 0.001, Miettinen & Nurminen; Difference in Percentage = 40.4, 95% CI 2-sided [19.6 to 57.0]

7. Primary Outcome: Percentage of Participants With a Systemic Adverse Event Prompted on the Vaccination Report Card
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the study vaccine. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an AE. VRC-prompted systemic AEs included non-injection-site varicella-like and herpes zoster (HZ)-like rashes. The percentage of participants with one or more VRC-prompted systemic AE was assessed with incidence > 0% in one or more vaccination groups.
Time Frame: Up to ~28 days Postdose 4 (Up to ~118 days)
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1: Heat-treated Varicella-Zoster Virus (VZV) Vaccine | Part 1: Gamma-Irradiated VZV Vaccine A | Part 1: Placebo | Part 2: Gamma-Irradiated VZV Vaccine B | Part 2: Gamma-Irradiated VZV Vaccine C
Number analyzed (Participants) | 64 | 61 | 32 | 63 | 65
Percentage of Participants | 45.3 | 54.1 | 50.0 | 52.4 | 41.5
Statistical Analysis 1: Comparison: Part 1: Heat-treated Varicella-Zoster Virus (VZV) Vaccine vs Part 1: Placebo; Test type: Other; Difference in Percentage = -4.7, 95% CI 2-sided [-25.3 to 16.1] — Miettinen & Nurminen
Statistical Analysis 2: Comparison: Part 1: Gamma-Irradiated VZV Vaccine A vs Part 1: Placebo; Test type: Other; Difference in Percentage = 4.1, 95% CI 2-sided [-16.9 to 24.9] — Miettinen & Nurminen

8. Primary Outcome: Percentage of Participants With Elevated Temperature Prompted on the Vaccination Report Card
Description: Elevated temperature is defined as ≥100.5 °F (≥38.1 °C), oral equivalent. The percentage of participants with VRC-prompted elevated temperature was assessed.
Time Frame: Up to ~28 days Postdose 4 (Up to ~118 days)
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1: Heat-treated Varicella-Zoster Virus (VZV) Vaccine | Part 1: Gamma-Irradiated VZV Vaccine A | Part 1: Placebo | Part 2: Gamma-Irradiated VZV Vaccine B | Part 2: Gamma-Irradiated VZV Vaccine C
Number analyzed (Participants) | 64 | 61 | 32 | 63 | 65
Percentage of Participants | 1.6 | 1.6 | 0.0 | 3.2 | 1.5
Statistical Analysis 1: Comparison: Part 1: Heat-treated Varicella-Zoster Virus (VZV) Vaccine vs Part 1: Placebo; Test type: Other; p = 0.480, Miettinen & Nurminen; Difference in Percentage = 1.6, 95% CI 2-sided [-9.3 to 8.4]
Statistical Analysis 2: Comparison: Part 1: Gamma-Irradiated VZV Vaccine A vs Part 1: Placebo; Test type: Other; p = 0.469, Miettinen & Nurminen; Difference in Percentage = 1.6, 95% CI 2-sided [-9.2 to 8.8]

9. Primary Outcome: Percentage of Participants Who Discontinued the Study Drug Due to an Adverse Event
Description: An adverse event (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the study vaccine. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an AE. The percentage of participants who discontinued the study drug due to one or more AEs was assessed.
Time Frame: Up to Dose 4 (Up to ~90 days)
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1: Heat-treated Varicella-Zoster Virus (VZV) Vaccine | Part 1: Gamma-Irradiated VZV Vaccine A | Part 1: Placebo | Part 2: Gamma-Irradiated VZV Vaccine B | Part 2: Gamma-Irradiated VZV Vaccine C
Number analyzed (Participants) | 64 | 61 | 32 | 63 | 65
Percentage of Participants | 0.0 | 0.0 | 0.0 | 1.6 | 0.0
Statistical Analysis 1: Comparison: Part 1: Heat-treated Varicella-Zoster Virus (VZV) Vaccine vs Part 1: Placebo; Test type: Other; Difference in Percentage = 0.0, 95% CI 2-sided [-10.8 to 5.7] — Miettinen & Nurminen
Statistical Analysis 2: Comparison: Part 1: Gamma-Irradiated VZV Vaccine A vs Part 1: Placebo; Test type: Other; Difference in Percentage = 0.0, 95% CI 2-sided [-10.8 to 6.0] — Miettinen & Nurminen

ADVERSE EVENTS:
Time Frame: Up to ~28 days Postdose 4 (up to ~118 days)
Description: All participants who received at least one dose of vaccine and who had any safety follow-up were included in the safety evaluation, based on the actual vaccination received. Participants were excluded from the safety analysis population if they received an incorrect vaccination.
Groups:
- Part 1 Heat-treated VZV Vaccine; Gamma-irradiated VZV Vaccine A; Part 2 Gamma-irradiated VZV Vaccine B; Gamma-irradiated VZV Vaccine C: Participants received an 0.65 mL subcutaneous injection of heat-treated varicella zoster virus (VZV) vaccine or alternative inactivation method VZV vaccine A, B, C; 4-dose regimen administered ~30 days apart.
- Placebo: Participants received a 4-dose placebo regimen administered ~30 days apart.
Arm/Group | Part 1 Heat-treated VZV Vaccine | Gamma-irradiated VZV Vaccine A | Placebo | Part 2 Gamma-irradiated VZV Vaccine B | Gamma-irradiated VZV Vaccine C
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/61 | 0/32 | 0/63 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/64 | 1/61 | 0/32 | 1/63 | 0/65
Other Adverse Events (participants affected / at risk) | 47/64 | 48/61 | 20/32 | 47/63 | 43/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Heat-treated VZV Vaccine (N=64) | Gamma-irradiated VZV Vaccine A (N=61) | Placebo (N=32) | Part 2 Gamma-irradiated VZV Vaccine B (N=63) | Gamma-irradiated VZV Vaccine C (N=65)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Heat-treated VZV Vaccine (N=64) | Gamma-irradiated VZV Vaccine A (N=61) | Placebo (N=32) | Part 2 Gamma-irradiated VZV Vaccine B (N=63) | Gamma-irradiated VZV Vaccine C (N=65)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye allergy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scleral disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (4) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 29 (73) | 31 (73) | 2 (2) | 28 (69) | 27 (73)
Injection site haematoma (General disorders) | 4 (4) | 5 (6) | 1 (1) | 5 (5) | 1 (1)
Injection site induration (General disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Injection site pain (General disorders) | 32 (80) | 36 (79) | 7 (7) | 40 (86) | 32 (73)
Injection site papule (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 10 (13) | 7 (12) | 0 (0) | 7 (11) | 5 (8)
Injection site rash (General disorders) | 2 (2) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 29 (66) | 20 (42) | 3 (3) | 24 (53) | 24 (60)
Injection site warmth (General disorders) | 4 (4) | 1 (2) | 0 (0) | 4 (4) | 3 (3)
Local swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 3 (3) | 2 (4) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (5) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bed bug infestation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 3 (3) | 1 (2) | 1 (1) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (4) | 5 (6) | 3 (3) | 0 (0) | 3 (3)
Oral herpes (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 3 (3) | 3 (3) | 2 (4) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 4 (4) | 1 (1) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (5)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5) | 0 (0) | 3 (4) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (9) | 1 (2) | 0 (0) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (10) | 6 (9) | 3 (3) | 9 (19) | 8 (19)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Generalised anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (5) | 1 (1)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (7)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (3) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Heat rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 4 (6) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 2 (3)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash vesicular (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.